CLINICAL TRIAL: NCT03425175
Title: Audio Recording During Laparoscopic Surgery - The Impact on Conversation Between Surgeons
Brief Title: Audio Recording During Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Erik Stenberg, MD, PhD, Principal Investigator, Region Örebro County
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EPN 2017/247
Record Dates: First submitted 2018-01-24; First posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Perioperative/Postoperative Complications; Laparoscopy; Communication; Communication, Multidisciplinary
Keywords: Non-relevant conversation; Surgical safety; Audio recording
MeSH Terms: conditions — Postoperative Complications; Communication

STUDY DESIGN:
Intervention Model Description: Non-randomised intervenion
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Standard care with recording of video but no audio-recording
- Intervention group (Experimental): Standard care with the addition of simultaneous audio-recording during the operation.
  Interventions: Other: Audio-recoring

INTERVENTIONS:
Other: Audio-recoring — Recording of audio through microphone carried bu surgeon and assistant surgeon
  Arms: Intervention group

SUMMARY:
In september 2017 audio recording during laparoscopic general surgery was implemented as routine a Lindesbergs hospital. The study was designed to observe operations before and after the introduction of audio recording. The main outcome of the study was time spent on non-relevant conversation.

DETAILED DESCRIPTION:
In september 2017 audio recording during laparoscopic general surgery was implemented as routine a Lindesbergs hospital. One single observer not working at the department observed consecutive operations before and after the introduction of audio recordings. All elective laparoscopic procedures were included. There was no available data to support a Power-calculation why we intended to include 20 patients in each arm of the study. Exclusion criteria were refusal of operating team or patient to participate in the study, or planned open surgery. Potential disturbances were recorded by the observer. The main outcome was time with non-relevant conversation (for the operation or as part of education).

ELIGIBILITY:
Inclusion Criteria: Elective laparoscopic general surgery -

Exclusion Criteria:R, planned open surgery, refusal to participate (patient or operating team)

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Non-relevant conversation | Operation. Measured from from the start of the operation (WHO surgical safety checklist) until end of operation (last stitch in place)
  Time spent on non-relevant conversation

SECONDARY OUTCOMES:
Postoperative complication | 30 days after surgery
  complication occuring within the first 30 Days after surgery
Intraoperative unplanned event | Operation. Measured from from the start of the operation (WHO surgical safety checklist) until end of operation (last stitch in place)
  Any deviation from expected events during the surgical procedure
Corrections of assistant surgeon | Operation. Measured from from the start of the operation (WHO surgical safety checklist) until end of operation (last stitch in place)
  number of corrections of assistant surgeon made by the operating surgeon
Operation time | Operation. Measured from from the start of the operation (WHO surgical safety checklist) until end of operation (last stitch in place)
  Length of operation

CONTACTS AND LOCATIONS:
Overall Officials: Erik Stenberg, MD, PhD, Principal Investigator — Örebro University, Region Örebro Län
Locations (1):
- Lindesbergs Hospital, Lindesberg, Sweden

IPD SHARING:
Plan to Share IPD: No
All results

REFERENCES:
- [Derived] Bergstrom H, Larsson LG, Stenberg E. Audio-video recording during laparoscopic surgery reduces irrelevant conversation between surgeons: a cohort study. BMC Surg. 2018 Nov 6;18(1):92. doi: 10.1186/s12893-018-0428-x. PMID 30400860